CLINICAL TRIAL: NCT00206310
Title: Controlled Rosuvastatin Multinational Study in Heart Failure CORONA A Randomized, Double-Blind, Placebo Controlled Phase III Study With Rosuvastatin in Subjects With Chronic Symptomatic Systolic Heart Failure
Brief Title: Crestor Versus Placebo in Subjects With Heart Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4522IL/0098; D3562C00098; CORONA
Record Dates: First submitted 2005-09-16; First posted 2005-09-21 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: CRESTOR

SUMMARY:
The purpose of the study is to investigate if rosuvastatin, added on top of all other medicines prescribed to subjects with symptomatic systolic heart failure, reduces the combined endpoint of cardiovascular death or non-fatal myocardial infarction or non-fatal stroke (time to first event)

ELIGIBILITY:
Inclusion Criteria:

* Chronic symptomatic systolic heart failure of ischaemic aetiology as judged by the investigator, optimal therapy for chronic symptomatic systolic heart failure according to the investigator

Exclusion Criteria:

* Acute myocardial infarction within 6 months before randomization
* Treatment with any statin or other lipid lowering drug; or a medical condition that in the opinion of the investigator requires treatment with a statin or other lipid lowering drug

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5013
Dates: Start 2003-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether rosuvastatin reduces the combined endpoint of cardiovascular death or non-fatal myocardial infarction (MI) or non-fatal stroke (time to first event).

SECONDARY OUTCOMES:
The secondary objectives are to evaluate the effects of rosuvastatin on:
Total mortality
Any coronary event defined as the combined endpoint of sudden death or fatal or non-fatal MI or Percutaneous Transluminal Coronary Angioplasty (PTCA) or Coronary Artery Bypass Grafting (CABG) or defibrillation of ventricular fibrillation by an implant
Cardiovascular mortality with cause-specific mortality for sudden death; fatal MI; and death from worsening heart failure
Total number of hospitalizations for cardiovascular causes; for unstable angina; and for worsening heart failure

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Medical Science Director, MD, Study Director — AstraZeneca
Locations (375):
- Belgium (13):
  - Research Site, Aalst
  - Research Site, Bouge
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Ensival
  - Research Site, Fléron
  - Research Site, Genk
  - Research Site, Huy
  - Research Site, Leuven
  - Research Site, Mol
  - Research Site, Turnhout
  - Research Site, Verviers
- Bulgaria (5):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Czechia (21):
  - Research Site, Bene¿ov U Prahy
  - Research Site, Bene¿ov
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Hradec Králové 5
  - Research Site, Jihlava
  - Research Site, Kladno
  - Research Site, Liberec
  - Research Site, Ostrava
  - Research Site, Ostrava 3 - Vítkovice
  - Research Site, Pelh¿imov
  - Research Site, Plze¿-Bory
  - Research Site, Plze¿
  - Research Site, Prague
  - Research Site, P¿íbram V - Zdabo¿
  - Research Site, P¿íbram
  - Research Site, Slaný
  - Research Site, Tábor
  - Research Site, Ústí nad Labem
  - Research Site, ¿eská Lípa
  - Research Site, ¿eské Bud¿jovice
- Denmark (19):
  - Research Site, Aalborg
  - Research Site, Copenhagen
  - Research Site, Elsinore
  - Research Site, Esbjerg
  - Research Site, Frederiksberg
  - Research Site, Frederikssund
  - Research Site, Glostrup Municipality
  - Research Site, Haderslev
  - Research Site, Horsens
  - Research Site, Hvidovre
  - Research Site, Kbh. S
  - Research Site, Kolding
  - Research Site, København N
  - Research Site, København Ø
  - Research Site, Næstved
  - Research Site, Odense C
  - Research Site, Roskilde
  - Research Site, Svendborg
  - Research Site, Viborg
- Finland (13):
  - Research Site, Helsinki
  - Research Site, Hyvinkää
  - Research Site, Jakobstad
  - Research Site, Kemi
  - Research Site, Kokkola
  - Research Site, Lahti
  - Research Site, Lappeenranta
  - Research Site, Mariehamn
  - Research Site, Oulu
  - Research Site, Porvoo
  - Research Site, Seinäjoki
  - Research Site, Tampere
  - Research Site, Uusikaupunki
- France (28):
  - Research Site, Allauch
  - Research Site, Antony
  - Research Site, Arras
  - Research Site, Cambrai
  - Research Site, Cergy-Pontoise
  - Research Site, Chambray-lès-Tours
  - Research Site, Chantepie
  - Research Site, Cholet
  - Research Site, Croix
  - Research Site, Dechy
  - Research Site, Gonesse
  - Research Site, Grenoble
  - Research Site, Le Coudray
  - Research Site, Lille
  - Research Site, Montfermeil
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Roubaix
  - Research Site, Saint-Denis
  - Research Site, Saint-Herblain
  - Research Site, Salouël
  - Research Site, Senlis
  - Research Site, Six-Fours-les-Plages
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Valenciennes
- Germany (56):
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, München, Bavaria
  - Research Site, Regensburg, Bavaria
  - Research Site, Cottbus, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Frankfurt am Main, Hesse
  - Research Site, Göttingen, Lower Saxony
  - Research Site, Hanover, Lower Saxony
  - Research Site, Greifswald, Mecklenburg-Vorpommern
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Saarbrücken, Saarland
  - Research Site, Dresden, Saxony
  - Research Site, Leipzig, Saxony
  - Research Site, Halle, Saxony-Anhalt
  - Research Site, Bad Segeberg, Schleswig-Holstein
  - Research Site, Lübeck, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
  - Research Site, Jena-Maua, Thuringia
  - Research Site, Aachen
  - Research Site, Bad Nauheim
  - Research Site, Bad Neustadt an der Saale
  - Research Site, Bad Wörishofen
  - Research Site, Berlin
  - Research Site, Brandenburg
  - Research Site, Braunschweig
  - Research Site, Coburg
  - Research Site, Cottbus
  - Research Site, Dillingen
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Görlitz
  - Research Site, Göttingen
  - Research Site, Greifswald
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Kassel
  - Research Site, Leipzig
  - Research Site, Leisnig
  - Research Site, Löbau
  - Research Site, Lübeck
  - Research Site, Mannheim
  - Research Site, München
  - Research Site, Neustadt/Aisch
  - Research Site, Norderstedt
  - Research Site, Nordhorn
  - Research Site, Regensburg
  - Research Site, Riesa
  - Research Site, Rüdersdorf
  - Research Site, Timmendorfer Strand
  - Research Site, Tübingen
  - Research Site, Vechta
  - Research Site, Wedel
  - Research Site, Wermsdorf
  - Research Site, Wolmirstedt
- Hungary (12):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Mosonmagyaróvár
  - Research Site, Sopron
  - Research Site, Szentes
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
- Ireland (3):
  - Research Site, Ballinasloe, Co. Galway
  - Research Site, Dublin
  - Research Site, Ryhope, Sunderland
- Netherlands (48):
  - Research Site, 's-Hertogenbosch
  - Research Site, Alkmaar
  - Research Site, Almelo
  - Research Site, Amersfoort
  - Research Site, Amsterdam
  - Research Site, Apeldoorn
  - Research Site, Blaricum
  - Research Site, Breda
  - Research Site, Capelle aan den IJssel
  - Research Site, Delft
  - Research Site, Den Helder
  - Research Site, Deventer
  - Research Site, Dirksland
  - Research Site, Dordrecht
  - Research Site, Ede
  - Research Site, Enschede
  - Research Site, Goes
  - Research Site, Gorinchem
  - Research Site, Gouda
  - Research Site, Groningen
  - Research Site, Haarlem
  - Research Site, Hardenberg
  - Research Site, Heerenveen
  - Research Site, Heerlen
  - Research Site, Helmond
  - Research Site, Hengelo
  - Research Site, Hilversum
  - Research Site, Hoofddorp
  - Research Site, Leiden
  - Research Site, Lelystad
  - Research Site, Maastricht
  - Research Site, Nijmegen
  - Research Site, Oss
  - Research Site, Roermond
  - Research Site, Roosendaal
  - Research Site, Rotterdam
  - Research Site, Schiedam
  - Research Site, Sittard
  - Research Site, Sneek
  - Research Site, The Hague
  - Research Site, Tiel
  - Research Site, Tilburg
  - Research Site, Veldhoven
  - Research Site, Velp
  - Research Site, Venlo
  - Research Site, Zeist
  - Research Site, Zoetermeer
  - Research Site, Zwolle
- Norway (12):
  - Research Site, Arendal
  - Research Site, Drammen
  - Research Site, Flekkefjord
  - Research Site, Fredrikstad
  - Research Site, Førde
  - Research Site, Gjettum
  - Research Site, Gjøvik
  - Research Site, Hamar
  - Research Site, Lillehammer
  - Research Site, Oslo
  - Research Site, Porsgrunn
  - Research Site, Tromsø
- Poland (27):
  - Research Site, Bialystok
  - Research Site, Bia¿ystok
  - Research Site, Bydgoszcz
  - Research Site, Chojnice
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Gliwice
  - Research Site, Inowroc¿aw
  - Research Site, I¿awa
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Ostrowiec ¿wi¿tokrzyski
  - Research Site, O¿awa
  - Research Site, Piotrkow Trybunalski
  - Research Site, Poznan
  - Research Site, Ruda ¿l¿ska
  - Research Site, Siedlce
  - Research Site, Skierniewice
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zamo¿¿
  - Research Site, ¿ód¿
  - Research Site, ¿yrardów
- Portugal (10):
  - Research Site, Almada
  - Research Site, Amadora
  - Research Site, Barreiro
  - Research Site, Carnaxide
  - Research Site, Coimbra
  - Research Site, Funchal
  - Research Site, Lisbon
  - Research Site, Penafiel
  - Research Site, Porto
  - Research Site, Vila Franca de Xira
- Romania (5):
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Craiova
  - Research Site, Târgu Mureş
- Research Site, Moscow, Russia, Russia
- Slovakia (9):
  - Research Site, Bardejov
  - Research Site, Bratislava
  - Research Site, Dolný Kubín
  - Research Site, Ko¿ice
  - Research Site, Lu¿enec
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Pre¿ov
  - Research Site, Rimavská Sobota
- South Africa (9):
  - Research Site, Bloemfontein, Free State
  - Research Site, Soweto, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Somerset West, Western Cape
  - Research Site, Bloemfontein
  - Research Site, Cape Town
  - Research Site, Lyttelton Manor
  - Research Site, Parktown
  - Research Site, Tygerberg
- Spain (18):
  - Research Site, Santiago, A Coruña
  - Research Site, Santiago de Compostela, A Coruña
  - Research Site, San Juan, Alicante
  - Research Site, Badalona, Barcelona
  - Research Site, Barcelona, Barcelona
  - Research Site, Terrassa, Barcelona
  - Research Site, Santander, Cantabria
  - Research Site, Castellon, Castellón
  - Research Site, A Coruña, Galicia
  - Research Site, San Sebastián, Guipuzcoa
  - Research Site, Alcorcón, Madrid
  - Research Site, Madrid, Madrid
  - Research Site, Marbella, Málaga
  - Research Site, Málaga, Málaga
  - Research Site, Palma de Mallorca, Palma de Mallorca
  - Research Site, Vigo, Pontevedra
  - Research Site, Salamanca, Salamanca
  - Research Site, Seville, Sevilla
- Sweden (16):
  - Research Site, Ängelholm
  - Research Site, Danderyd
  - Research Site, Eksjö
  - Research Site, Enköping
  - Research Site, Gothenburg
  - Research Site, Hudiksvall
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Linköping
  - Research Site, Lund
  - Research Site, Motala
  - Research Site, Mölndal
  - Research Site, Oskarshamn
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västervik
- Switzerland (6):
  - Research Site, Bellinzona
  - Research Site, Bern
  - Research Site, Geneva
  - Research Site, Lugano
  - Research Site, Schlieren
  - Research Site, Zurich
- United Kingdom (44):
  - Research Site, Cottingham, Hull
  - Research Site, Sidcup, Kent
  - Research Site, Airdrie, Lanarkshire
  - Research Site, Essex, London
  - Research Site, Antrim, Northern Ireland
  - Research Site, Belfast, Northern Ireland
  - Research Site, Paisley, Renfrewhsire
  - Research Site, Bridgend, Wales
  - Research Site, Aberdeen
  - Research Site, Ayr
  - Research Site, Basingstoke
  - Research Site, Belfast
  - Research Site, Blackpool
  - Research Site, Bridgend
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, Carshalton
  - Research Site, Croyden
  - Research Site, Croydon
  - Research Site, Durham
  - Research Site, East Kilbride
  - Research Site, Edinburgh
  - Research Site, Essex
  - Research Site, Glasgow
  - Research Site, Hastings
  - Research Site, High Wycombe
  - Research Site, Hull
  - Research Site, Kent
  - Research Site, Kirkcaldy
  - Research Site, Leicester
  - Research Site, Liverpool
  - Research Site, Llantrisant
  - Research Site, London
  - Research Site, Middlesex
  - Research Site, Newport
  - Research Site, Northumberland
  - Research Site, Paisley
  - Research Site, Poole
  - Research Site, Ryhope, Sunderland
  - Research Site, Scunthorpe
  - Research Site, Sheffield
  - Research Site, Sunderland
  - Research Site, West Bromwich
  - Research Site, York

REFERENCES:
- [Derived] Askevold ET, Gullestad L, Nymo S, Kjekshus J, Yndestad A, Latini R, Cleland JG, McMurray JJ, Aukrust P, Ueland T. Secreted Frizzled Related Protein 3 in Chronic Heart Failure: Analysis from the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA). PLoS One. 2015 Aug 19;10(8):e0133970. doi: 10.1371/journal.pone.0133970. eCollection 2015. PMID 26288364
- [Derived] Perez AC, Jhund PS, Stott DJ, Gullestad L, Cleland JG, van Veldhuisen DJ, Wikstrand J, Kjekshus J, McMurray JJ. Thyroid-stimulating hormone and clinical outcomes: the CORONA trial (controlled rosuvastatin multinational study in heart failure). JACC Heart Fail. 2014 Feb;2(1):35-40. doi: 10.1016/j.jchf.2013.07.008. Epub 2014 Jan 25. PMID 24622117
- [Derived] Gravning J, Askevold ET, Nymo SH, Ueland T, Wikstrand J, McMurray JJ, Aukrust P, Gullestad L, Kjekshus J; CORONA Study Group. Prognostic effect of high-sensitive troponin T assessment in elderly patients with chronic heart failure: results from the CORONA trial. Circ Heart Fail. 2014 Jan;7(1):96-103. doi: 10.1161/CIRCHEARTFAILURE.113.000450. Epub 2013 Nov 27. PMID 24284025
- [Derived] Perez AC, Jhund P, Preiss D, Kjekshus J, McMurray JJ. Effect of rosuvastatin on fatigue in patients with heart failure. J Am Coll Cardiol. 2013 Mar 12;61(10):1121-2. doi: 10.1016/j.jacc.2012.12.004. No abstract available. PMID 23473415
- [Derived] van der Velde AR, Gullestad L, Ueland T, Aukrust P, Guo Y, Adourian A, Muntendam P, van Veldhuisen DJ, de Boer RA. Prognostic value of changes in galectin-3 levels over time in patients with heart failure: data from CORONA and COACH. Circ Heart Fail. 2013 Mar;6(2):219-26. doi: 10.1161/CIRCHEARTFAILURE.112.000129. Epub 2013 Feb 8. PMID 23395934
- [Derived] Askevold ET, Nymo S, Ueland T, Gravning J, Wergeland R, Kjekshus J, Yndestad A, Cleland JG, McMurray JJ, Aukrust P, Gullestad L. Soluble glycoprotein 130 predicts fatal outcomes in chronic heart failure: analysis from the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA). Circ Heart Fail. 2013 Jan;6(1):91-8. doi: 10.1161/CIRCHEARTFAILURE.112.972653. Epub 2012 Dec 10. PMID 23230311
- [Derived] Gullestad L, Ueland T, Kjekshus J, Nymo SH, Hulthe J, Muntendam P, McMurray JJ, Wikstrand J, Aukrust P. The predictive value of galectin-3 for mortality and cardiovascular events in the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA). Am Heart J. 2012 Dec;164(6):878-83. doi: 10.1016/j.ahj.2012.08.021. Epub 2012 Oct 29. PMID 23194488
- [Derived] Latini R, Gullestad L, Masson S, Nymo SH, Ueland T, Cuccovillo I, Vardal M, Bottazzi B, Mantovani A, Lucci D, Masuda N, Sudo Y, Wikstrand J, Tognoni G, Aukrust P, Tavazzi L; Investigators of the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA) and GISSI-Heart Failure (GISSI-HF) trials. Pentraxin-3 in chronic heart failure: the CORONA and GISSI-HF trials. Eur J Heart Fail. 2012 Sep;14(9):992-9. doi: 10.1093/eurjhf/hfs092. Epub 2012 Jun 27. PMID 22740508
- [Derived] Stein EA, Vidt DG, Shepherd J, Cain VA, Anzalone D, Cressman MD. Renal safety of intensive cholesterol-lowering treatment with rosuvastatin: a retrospective analysis of renal adverse events among 40,600 participants in the rosuvastatin clinical development program. Atherosclerosis. 2012 Apr;221(2):471-7. doi: 10.1016/j.atherosclerosis.2011.12.011. Epub 2012 Jan 3. PMID 22304793
- [Derived] Ueland T, Dahl CP, Kjekshus J, Hulthe J, Bohm M, Mach F, Goudev A, Lindberg M, Wikstrand J, Aukrust P, Gullestad L. Osteoprotegerin predicts progression of chronic heart failure: results from CORONA. Circ Heart Fail. 2011 Mar;4(2):145-52. doi: 10.1161/CIRCHEARTFAILURE.110.957332. Epub 2011 Jan 7. PMID 21216833
- [Derived] McMurray JJ, Dunselman P, Wedel H, Cleland JG, Lindberg M, Hjalmarson A, Kjekshus J, Waagstein F, Apetrei E, Barrios V, Bohm M, Kamensky G, Komajda M, Mareev V, Wikstrand J; CORONA Study Group. Coenzyme Q10, rosuvastatin, and clinical outcomes in heart failure: a pre-specified substudy of CORONA (controlled rosuvastatin multinational study in heart failure). J Am Coll Cardiol. 2010 Oct 5;56(15):1196-204. doi: 10.1016/j.jacc.2010.02.075. PMID 20883926
- [Derived] Inglis SC, McMurray JJ, Bohm M, Schaufelberger M, van Veldhuisen DJ, Lindberg M, Dunselman P, Hjalmarson A, Kjekshus J, Waagstein F, Wedel H, Wikstrand J; CORONA Study Group. Intermittent claudication as a predictor of outcome in patients with ischaemic systolic heart failure: analysis of the Controlled Rosuvastatin Multinational Trial in Heart Failure trial (CORONA). Eur J Heart Fail. 2010 Jul;12(7):698-705. doi: 10.1093/eurjhf/hfq070. Epub 2010 May 25. PMID 20501489
- [Derived] McMurray JJ, Kjekshus J, Gullestad L, Dunselman P, Hjalmarson A, Wedel H, Lindberg M, Waagstein F, Grande P, Hradec J, Kamensky G, Korewicki J, Kuusi T, Mach F, Ranjith N, Wikstrand J; CORONA Study Group. Effects of statin therapy according to plasma high-sensitivity C-reactive protein concentration in the Controlled Rosuvastatin Multinational Trial in Heart Failure (CORONA): a retrospective analysis. Circulation. 2009 Dec 1;120(22):2188-96. doi: 10.1161/CIRCULATIONAHA.109.849117. Epub 2009 Nov 16. PMID 19917888
- [Derived] Kjekshus J, Apetrei E, Barrios V, Bohm M, Cleland JG, Cornel JH, Dunselman P, Fonseca C, Goudev A, Grande P, Gullestad L, Hjalmarson A, Hradec J, Janosi A, Kamensky G, Komajda M, Korewicki J, Kuusi T, Mach F, Mareev V, McMurray JJ, Ranjith N, Schaufelberger M, Vanhaecke J, van Veldhuisen DJ, Waagstein F, Wedel H, Wikstrand J; CORONA Group. Rosuvastatin in older patients with systolic heart failure. N Engl J Med. 2007 Nov 29;357(22):2248-61. doi: 10.1056/NEJMoa0706201. Epub 2007 Nov 5. PMID 17984166